CLINICAL TRIAL: NCT00345280
Title: Chosen Parameters of the Immune Response in the Origin of Ocular Changes in Patients With Cystic Fibrosis
Brief Title: Ocular Surface Changes in Patients With Cystic Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Bialystok (Other Government)
Responsible Party: Malgorzata Mrugacz, Medical University of Bialystok, Poland
Other Study IDs: 8789; N40605131/1894
Record Dates: First submitted 2006-06-27; First posted 2006-06-28 (Estimated); Last update posted 2008-06-17 (Estimated); Status verified 2008-06

CONDITIONS: Eye Manifestations
Keywords: Cystic fibrosis; eye; inflammation; apoptosis; C11+
MeSH Terms: conditions — Eye Manifestations; Cystic Fibrosis; Inflammation; Lipodystrophy, Congenital Generalized

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: impression cytology, obtain the tear fluid — Vitamin A
  Other Names: Becton Dickinson

SUMMARY:
Cystic fibrosis(CF) is an inherited disease affecting children, adolescents and young adults with dysfunction of secretory glands.It is caused by mutations in the protein-coding gene which function as the cystic fibrosis transmembrane regulator (CFTR), responsible for the secretion of chloride ions in epithelial cells, adenocytes, sweat gland cells, pancreatic ducts,alimentary and respiratory tracts and eye. Assessment of the relationship between the inflammatory processes and apoptosis in the eye in the course of cystic fibrosis will allow determination of immunological exponents which may facilitate diagnosis.

DETAILED DESCRIPTION:
The aim: To assess the role of chosen parameters of immunological response in the induction of ocular changes in cystic fibrosis patients, particularly chosen chemokine concentrations in the tear fluid and analysis of chosen apoptotic markers expression on conjunctival epithelial cells.

ELIGIBILITY:
Inclusion Criteria:

* male and female patients aged 3-25 with clinically definite diagnosis of cystic fibrosis
* all patients must give written consent for participation in the study at screening

Exclusion Criteria:

* patients with a history of chronic disease of the immune system
* patients with the history of systemic diseases
* patients with the history chronic ocular diseases
* patients who have been treated with corticosteroids in the past 3 months prior to the screening visit

Ages: 3 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: 26 male and female patients aged 3-25 with clinically definite diagnosis of cystic fibrosis
Sampling Method: Probability Sample
Enrollment: 26 (Estimated)
Dates: Start 2006-08; Study Completion 2008-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Mrugacz, MD, PhD, Principal Investigator — Department of Pediatric Ophthalmology Medical University of Bialystok, Poland
Locations (1):
- Medical University, Bialystok, Poland